CLINICAL TRIAL: NCT03831217
Title: Long Term Outcome Women Who Undergone Mid-urethral Sling Surgery Using Urogynecologic Ultrasonographic and Urodynamic Evaluation
Brief Title: Long Term Outcome Women Who Undergone Mid-urethral Sling Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, kaan baydemir, kaan baydemir md, Ankara University
Other Study IDs: 29081991
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2019-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Trans-Obturator Tape; Tension-Free Vaginal Tape; Mid-Urethral Sling surgeries; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mid urethral sling surgery — patients with clinically and/or urodynamically proven stress urinary incontinence underwent mid urethral sling surgery under general anesthesia.

SUMMARY:
The patients who underwent mid-urethral sling surgery for stress urinary incontinence will evaluate. The aim of our study is to assess long term surgical outcomes and post operative clinical findings include physical examinations, quality of life questionnaires, ultrasonographic measurements.

DETAILED DESCRIPTION:
Patients who underwent mid-urethral sling surgery in Ankara University Obstetrics and Gynecology Department since 2007 will be included.

Primary outcome measure is to describe factors effecting long term success in mid-urethral sling surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery in Ankara University Obstetrics and Gynecology Department since 2007
* Patients come to follow up

Exclusion Criteria:

* inability in verbal and written communication
* impairment in cognitive functions

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients with underwent mid-urethral surgery in Ankara University Obstetrics and Gynecology Department since 2007 at any age.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Objective cure rates | 1-11 years
  Objective cure is negative cough stress test.
Subjective cure rates | 1-11 years
  Subjective cure is evaluated with PGI-I instrument. Patients who give 'much better' or 'better' response to the PGI question are considered subjectively cured.

SECONDARY OUTCOMES:
Tape localization | 1-11 years
  Length of urethra, length of mesh, distance between urethra and mesh, distance between mesh and bladder neck will be measured. The correlation between these parameters and surgical success will be evaluated
Quality of life(QoL) after surgery | 1-11 years
  Impact of surgery on quality of life will be evaluated by QoL questionnaire
Patient satisfaction | 1-11 years
  Patient satisfaction will be assessed using a 10-points Visual Analogue Scale (VAS) that ranged from ''complete achievement of my goal'' (10 points) to ''no achievement of my goal'' (0 points). Patient Global Impression of Improvement (PGI-I) and VAS scale correlation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaan Baydemir, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided